CLINICAL TRIAL: NCT04688359
Title: Nurse-coordinated Follow-up Program in Primary Care: a Mixed-method Complex Intervention Feasibility and RCT Pilot Trial Among People at Risk for T2DM.
Brief Title: Effectiveness of Nurse-coordinated Follow-up Program in Primary Care for People at Risk for T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Akureyri (Other)
Collaborators: Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UAkureyri
Record Dates: First submitted 2020-12-01; First posted 2020-12-30 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pre-diabetes; Cardiovascular Risk Factor; T2DM (Type 2 Diabetes Mellitus); Primary Health Care
Keywords: Pre-diabetes; Cardiovascular Risk Factors; Guided Self Determination; Intervention; Primary Health Care
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 2 groups one intervention group and one control group
Who Masked: Participant
Masking Description: The participants is informed of two groups but not which group he is allocated in.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Those receiving nurse-lead Guided Self Determination (GSD) for one to three times over six months starting four to six months after recruitment and first measurement.
  Interventions: Behavioral: Guided Self Determination
- Control group (No Intervention): Those not receiving nurse-lead Guided Self Determination (GSD) for one to three times over six months starting four to six months after recruitment and first measurement.

INTERVENTIONS:
Behavioral: Guided Self Determination — Nurse lead intervention in primary care
  Other Names: GSD
  Arms: Intervention group

SUMMARY:
Previous Icelandic studies regarding prevalence of diabetes have mostly used data from the capital area. Information on the proportion of people at risk at developing T2DM or having undiagnosed T2DM among people living in rural Northern Iceland is unknown. Clinical guidelines recommend that patients with prediabetes (diabetes warning signs) should be referred to a counselling program. The study will evaluate effectiveness of nurse-coordinated Guided Self-Determination (GSD) follow up program toward health promotion, for people at risk of T2DM.

DETAILED DESCRIPTION:
Prevalence of type 2 Diabetes Mellitus (T2DM) a major health problem is rising. This metabolic disease characterized by the inability to effectively metabolize glucose, and often also a silent and sneaky onset. A lag is often found between diagnose and onset of the disease. Diabetes related complications are expensive for the society, and reduce quality of life for the individual.

Around one out of three with T2DM in an Icelandic study were unaware of their T2DM when fasting blood glucose was measured. In the U.S.A., the average interval between onset of the disease and diagnose is seven years, and the authors claimed that 30% of people with T2DM are undiagnosed, with increased risk for chronic diabetes complications higher Cardiovascular risk factors (CVR), and higher premature death for people with early onset of T2DM compared to late onset of T2DM.

Research have shown 1.83-fold higher risk of CVD for those with prediabetes and 2.26-fold higher risk for individuals with undiagnosed diabetes compared to individuals with normal HbA1c. These results highlight the pivotal need to prevent development of diabetes, as there is an association between increased obesity and increased prevalence of T2DM as Type 2 diabetes (T2DM) is also found to be a major risk factor for cardiovascular diseases.

Icelandic people and especially men are becoming more overweight. From the years 1968-2012, body mass index (BMI) increased by 11%, from 25.8 kg/m2 to 28.7 kg/m2 for men between 50-69 years. In women 50-69 years, the BMI increased from 25.2 kg/m2 to 27.2 kg/m2, or 8%. These results highlight the pivotal need to prevent development of diabetes in Iceland, as there is an association between increased obesity and increased prevalence of type 2 Diabetes Mellitus (T2DM).

A Guided Self-Determination (GSD) is based on a strong theoretical value and is a well establish nurse-led interventional method for people diagnosed with T2DM and other diseases. To our knowledge this is the first time that GSD is used in Iceland. Nurses working in primary care, at The Health Care Institution of North Iceland (HSN), in Akureyri, Husavik and Sauðarkrokur, will offer the GSD intervention. Before the intervention the nurses will receive teaching and consultation from an experienced GSD diabetic nurse. During their use of the GSD method they will have counseling from the experienced GSD nurse and the PhD student. A systematic review claimed, that multi-professional interventions are more effective in improving diabetes care compared to single professional interventions.

A recent Cochrane review using data from 18 trials, investigated the impact of nurses working as substitutes for primary care doctors. The results demonstrate that using the capacity and skills of nurses to deliver primary healthcare services leads to similar or better patient health and higher patient satisfaction. As such, this might be an important strategy to improve access, efficiency, and quality of care, and at the same time strengthen health promotion aspects of care and management of chronic diseases and increase teamwork in primary care.

This study is a part of doctoral student study. This PhD project is collaboration between University of Akureyri, Iceland (UNAK), Western Norway University of Applied Sciences (HVL) and the Health Care Institution of North Iceland (HSN). HVL has a considerably experience in researching diabetes through the Diabetes Research Group for BEST Practice (DiaBEST). The research group DiaBEST consist of researchers from Bergen University Collage, the University of Bergen and the University of Stavanger. The projects contribute to increase knowledge about and implementation of evidence-based practice within primary care.

ELIGIBILITY:
Inclusion Criteria two of three:

* BMI ≥ 30 kg/m2,
* score ≥ 9 on FINDRISC,
* HbA1c level ≥ 42 mmol/mol.
* Non-blood-glucose-lowering medical treated T2DM.

Exclusion Criteria:

* People diagnosed with Diabetes at strart-point.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk Factors changes up to one year after an intervention | 0- 6 months and 1 year
  Changes for each participant from Baseline to endpoint on CVR factors, changes of risk measured in percentages (%) compared to normal risk in the Icelandic population from beginning to end of intervention. Using the Icelandic cardiovascular risk factor calculator.
Measurements behind the Icelandic heart association risk calculator | 0- 6 months and 1 year
  Changes from baseline to endpoint:
  * Weight and height (will be combined to report BMI in kg/m^2)
  * Systolic blood pressure: In mm hg
  * Cholesterol: in mmol/L
  * HDL-Cholesterol: in mmol/L
  * Triglycerides measurements: in mmol/L,
  * Regular physical activity: yes/no
  * Smoking: never, stopped, 1/2 pack or less a day, 1/2 to 1 pack a day, 1 pack or more
  * Do you have diabetes: yes/no,
  * Do gender parents, brothers or sisters of same parents, have cardiovascular diseases : Yes/No

SECONDARY OUTCOMES:
Changes in HbA1c level | 0- 6 months and 1 year
  Changes in HbA1c mmol/L, (normal less than 42 mmol/mol, prediabetes 42-48 mmol/mol, diabetes over 48 mmol/mol)
FINDRISC risk score "Diabetes Risk Score questionnaire" | 0- 6 months and 1 year
  Changes from beginning to end of intervention between groups score reported on a scale from 0 - 26, (normal under 9, increased risk 9 and over)
WHO-5 Quality of Life (QoL) questionnaire | 0- 6 months and 1 year
  Changes within and between groups from baseline to endpoint. Well-being index. The WHO-5 consists of five statements, which respondents rate according to the scale below (in relation to the past two weeks).
  marking x on 5 = All of the time marking x on 4 = Most of the time marking x on 3 = More than half of the time marking x on 2 = Less than half of the time marking x on 1 = Some of the time marking x on 0 = At no time The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
EQ-5D-5L Questionnaire of self rated health. | 0- 6 months and 1 year
  Changes from beginning to end of intervention within and between groups scoring from one to five at each of the five dimension 3125 definition of health state, Higher score worse outcome: Mobility dimension; Self-care dimension; Usual activities dimension; Pain/discomfort dimension; Anxiety/depression dimension.
  Respondents self-rate their level of severity for each dimension using five-levels:
  1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems 5 = unable to do/having extreme problems.
  Visual analogue scale; mark health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. At the both ends of the scale that the bottom rate (0) corresponds to " the worst health you can imagine", and the highest rate (100) "the best health you can imagine". higher score better outcome
Health Literacy (HL) questionnaire Icelandic version: HLS-EU-Q16IS. | 0- 6 months and 1 year
  Changes from beginning to end of intervention within and between groups 16 questions regarding health literacy. The Icelandic version asking the person from on the scale from; "very difficult", "fairly difficult", "fairly easy", "very easy",
  fairly easy and very easy are united into "easy" (scored with 1) very difficult, fairly difficult are united into "difficult" (scored with 0). score can range from 0 (low/no Health Literacy) to 16 (high Health Literacy)
  (Results will be grouped into two groups: less than 13 and over 13 points according to prior research results in Iceland)
Hip-to-Waist ratio | 0- 6 months and 1 year
  Changes from beginning to end of intervention in both groups Hip-to-Waist ratio measurement: cm/cm, increased risk if ratio over 1.0

OTHER OUTCOMES:
Changes in fastening glucose from start point to endpoint in both groups | 0- 6 months and 1 year
  Two hours fasting blood glucose level (2HFG): mmol/L,
LDL cholesterol changes from start point to endpoint in both groups | 0- 6 months and 1 year
  * LDL-Cholesterol:measured in mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Arun K Sigurdardottir, PhD, Study Director — University of Akureyri
Locations (1):
- University of Akureyri, Akureyri, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen K, Aspelund T, Gudmundsson EF, Siggeirsdottir K, Thorolfsdottir RB, Sigurdsson G, Gudnason V. [Five decades of coronary artery disease in Iceland. Data from the Icelandic Heart Association]. Laeknabladid. 2017 Oktober;103(10):411-420. doi: 10.17992/lbl.2017.10.153. Icelandic. PMID 29044036
- [Background] Kong AP, Luk AO, Chan JC. Detecting people at high risk of type 2 diabetes- How do we find them and who should be treated? Best Pract Res Clin Endocrinol Metab. 2016 Jun;30(3):345-55. doi: 10.1016/j.beem.2016.06.003. Epub 2016 Jun 11. PMID 27432070
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2016 Abridged for Primary Care Providers. Clin Diabetes. 2016 Jan;34(1):3-21. doi: 10.2337/diaclin.34.1.3. No abstract available. PMID 26807004
- [Background] Zoffmann V, Kirkevold M. Realizing empowerment in difficult diabetes care: a guided self-determination intervention. Qual Health Res. 2012 Jan;22(1):103-18. doi: 10.1177/1049732311420735. Epub 2011 Aug 29. PMID 21876206
- [Background] IDF.org,( 2017). International Diabetes Federation,Webside. About Diabetes.accessed 28th of June 2018
- [Background] Bahler C, Huber CA, Brungger B, Reich O. Multimorbidity, health care utilization and costs in an elderly community-dwelling population: a claims data based observational study. BMC Health Serv Res. 2015 Jan 22;15:23. doi: 10.1186/s12913-015-0698-2. PMID 25609174
- [Background] Thorsson B, Aspelund T, Harris TB, Launer LJ, Gudnason V. [Trends in body weight and diabetes in forty years in Iceland]. Laeknabladid. 2009 Apr;95(4):259-66. Icelandic. PMID 19420407
- [Background] Zhang Y, Hu G, Zhang L, Mayo R, Chen L. A novel testing model for opportunistic screening of pre-diabetes and diabetes among U.S. adults. PLoS One. 2015 Mar 19;10(3):e0120382. doi: 10.1371/journal.pone.0120382. eCollection 2015. PMID 25790106
- [Background] World Health Organization. (2018). Diabetes fact sheet. Available from: World Health Organization, web site: http: //www.who.int/mediacentre/factsheeds/fs312/en (accessed 28. June 2018)
- [Background] Saaristo T, Moilanen L, Jokelainen J, Korpi-Hyovalti E, Vanhala M, Saltevo J, Niskanen L, Peltonen M, Oksa H, Cederberg H, Tuomilehto J, Uusitupa M, Keinanen-Kiukaanniemi S. Cardiometabolic profile of people screened for high risk of type 2 diabetes in a national diabetes prevention programme (FIN-D2D). Prim Care Diabetes. 2010 Dec;4(4):231-9. doi: 10.1016/j.pcd.2010.05.005. Epub 2010 Jun 18. PMID 21134669
- [Background] Steinarsson AO, Rawshani A, Gudbjornsdottir S, Franzen S, Svensson AM, Sattar N. Short-term progression of cardiometabolic risk factors in relation to age at type 2 diabetes diagnosis: a longitudinal observational study of 100,606 individuals from the Swedish National Diabetes Register. Diabetologia. 2018 Mar;61(3):599-606. doi: 10.1007/s00125-017-4532-8. Epub 2018 Jan 9. PMID 29318343
- [Background] Laurant M, van der Biezen M, Wijers N, Watananirun K, Kontopantelis E, van Vught AJ. Nurses as substitutes for doctors in primary care. Cochrane Database Syst Rev. 2018 Jul 16;7(7):CD001271. doi: 10.1002/14651858.CD001271.pub3. PMID 30011347
- [Background] Gustafsdottir SS, Sigurdardottir AK, Arnadottir SA, Heimisson GT, Martensson L. Translation and cross-cultural adaptation of the European Health Literacy Survey Questionnaire, HLS-EU-Q16: the Icelandic version. BMC Public Health. 2020 Jan 14;20(1):61. doi: 10.1186/s12889-020-8162-6. PMID 31937293
- [Result] Seidu S, Walker NS, Bodicoat DH, Davies MJ, Khunti K. A systematic review of interventions targeting primary care or community based professionals on cardio-metabolic risk factor control in people with diabetes. Diabetes Res Clin Pract. 2016 Mar;113:1-13. doi: 10.1016/j.diabres.2016.01.022. Epub 2016 Jan 21. PMID 26972954
- [Derived] Arnardottir E, Sigurdardottir AK, Skinner T, Graue M, Kolltveit BH. Prediabetes and cardiovascular risk factors: the effectiveness of a guided self-determination counselling approach in primary health care, a randomized controlled trial. BMC Public Health. 2024 Nov 1;24(1):3035. doi: 10.1186/s12889-024-20538-1. PMID 39487428
- See also: Diabetes fact sheet 2018 — http://www.who.int/
- See also: International Diabetes Federation webside — http://idf.org